CLINICAL TRIAL: NCT02699112
Title: Improvement of Cardiac Function and Neural Respiratory Drive Following Set up of Non-invasive Ventilation in Patients With Hypercapnic Respiratory Failure Caused by Obesity Hypoventilation Syndrome
Brief Title: Cardiac and Respiratory Function With Non-invasive Ventilation
Acronym: CARE-NIV
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: University of Padova (Other); King's College London (Other); Lane Fox Respiratory (Other)
Responsible Party: Sponsor
Other Study IDs: 179324
Record Dates: First submitted 2016-01-27; First posted 2016-03-04 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: OHS; Hypercapnic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Parasternal EMG (EMGpara) and Transthoracic Echocardiography — OHS patients recruited will have EMGpara and Transthoracic Echocardiography at admission and when established on NIV at 3 months.

SUMMARY:
To assess patients with hypercapnic respiratory failure using echocardiography,cardiac output measurements and markers of neural respiratory drive (EMGpara) prior to, during and after non-invasive ventilation (NIV) initiation, and to follow the patients for 3 months. The investigators hypothesize that the improvement in cardiac function and/or respiratory mechanics over time are associated with ongoing improvements in oxygenation, quality of life and exercise capacity.

DETAILED DESCRIPTION:
Respiratory failure is characterized by the incapacity of the respiratory system to maintain the normal arterial blood gas homeostasis. Specifically, the overlap of hypoxaemia and hypercapnia (PaCO2 >6 kPa) is referred to as Hypercapnic Respiratory Failure (HRF). HRF is one of the most common causes for hospital admission with high re-admission rates, therefore constitute a major burden on healthcare systems. Non Invasive Ventilation (NIV) is a well established treatment in patients with hypercapnic respiratory failure who frequently suffer with associated pulmonary hypertension (PH). NIV helps to increase arterial oxygenation and reduces hypercapnia. It is used in patients with hypercapnic respiratory failure caused by Obesity Hypoventilation Syndrome (OHS). The associated degree of PH can lead to an increased afterload of the right ventricle (RV) that causes progressive remodelling of the right heart. RV dysfunction is correlated with a reduced long term prognosis in respiratory conditions. In literature NIV is shown as effective method to treat acute hypercapnic respiratory failure in OHS.

It has not been described how NIV impacts on cardiac function and NRD in OHS.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of OHS and Overlap Syndrome
* Hypercapnic respiratory failure with the need to commence NIV
* Expected to remain an inpatient for ≥ 24 hours
* Age ≥ 18 and <80 years
* BMI >30 kg/m2
* Confirmed sleep-disordered breathing
* Able to give informed consent to participation in the evaluation study
* Clinically stable without exacerbations for ≥ 6 weeks

Exclusion Criteria:

* Patients established on NIV
* Inability to tolerate NIV (< 4 hours usage at during hospital titration)
* Contraindication to NIV
* Requirement for immediate invasive mechanical ventilation at admission or any other acute critical illness
* Acute infective exacerbation
* Presence of other acute pathology or critical illness (such as pulmonary embolism)
* Presence of acute or chronic Left ventricular Cardiac Failure
* Significant Kidney or Liver disease
* Significant Anaemia
* History of Pulmonary Embolism in the previous 2 years
* Presence of cardiac congenital disease
* Presence of Primary Pulmonary Hypertension
* Presence of other severe medical problem, e.g. cancer and systemic connective tissue disease and vasculitides
* Pregnancy
* Psychological and social factors that would impair compliance with the evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with a confirmed diagnosis of OHS and Overlap Syndrome and hypercapnic respiratory failure with the clinical intervention to commence on NIV will be invited to participate in the trial.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Patients commencing on Non Invasive Ventilation (NIV); change in Cardiac Function from baseline and at 3 months | 3 months
  Patients with hypercapnic respiratory failure caused by obesity hypoventilation syndrome commencing on NIV; change in cardiac function using echocardiography at baseline and 3 months. Measurements taken prior to NIV initiation, and follow up at 3 months.
Patients commencing on Non Invasive Ventilation (NIV); change on Nueral Respiratory Drive (NRD) from baseline and at 3 months | 3 months
  Patients with hypercapnic respiratory failure caused by obesity hypoventilation syndrome commencing on NIV; change in markers of nerual respiratory drive/EMG para. Measurements taken prior to, and after NIV initiation, and follow up at 3 months.

SECONDARY OUTCOMES:
Patients commencing on Non Invasive Ventilation (NIV); change in Oxygenation from baseline, 6 weeks post initiation and at 3 months | 3 months
  To demonstrate that the improvement in cardiac function and/or respiratory mechanics over time are associated with ongoing improvements in oxygenation by taking samples of arterial blood gases.
  Measurements are made prior to, during and after NIV initiation, and follow up at 3 months.
Patients commencing on Non Invasive Ventilation (NIV); change in Quality of Life from baseline, 6 weeks post initiation and at 3 months | 3 months
  To demonstrate the hypothesis that the improvement in cardiac function and/or respiratory mechanics over time are associated with ongoing improvements in quality of life by asking participants to complete the Medical Research Council (MRC) dyspnoea scale. Measurement will be taken prior to NIV initiation, 6 weeks post initiation and at follow up at 3 months.
Patients commencing on Non Invasive Ventilation (NIV); change in Quality of Life from baseline, 6 weeks post initiation and at 3 months | 3 months
  To demonstrate the hypothesis that the improvement in cardiac function and/or respiratory mechanics over time are associated with ongoing improvements in quality of life by asking participants to complete the modified BORG Scale (breathlessness). Measurement will be taken prior to NIV initiation, 6 weeks post initiation and at follow up at 3 months.
Patients commencing on Non Invasive Ventilation (NIV); change in Quality of Life from baseline, 6 weeks post initiation and at 3 months | 3 months
  To demonstrate the hypothesis that the improvement in cardiac function and/or respiratory mechanics over time are associated with ongoing improvements in quality of life by asking participants to complete the St George's Respiratory Questionnaire (SGRQ). Measurement will be taken prior to NIV initiation, 6 weeks post initiation and at follow up at 3 months.
Patients commencing on Non Invasive Ventilation (NIV); change in Quality of Life from baseline, 6 weeks post initiation and at 3 months | 3 months
  To demonstrate the hypothesis that the improvement in cardiac function and/or respiratory mechanics over time are associated with ongoing improvements in quality of life by asking participants to complete the Hospital Anxiety and Depression Scale (HADS).
  Measurement will be taken prior to NIV initiation, 6 weeks post initiation and at follow up at 3 months.
Patients commencing on Non Invasive Ventilation (NIV); change in Quality of Life from baseline, 6 weeks post initiation and at 3 months | 3 months
  To demonstrate the hypothesis that the improvement in cardiac function and/or respiratory mechanics over time are associated with ongoing improvements in quality of life by asking participants to complete the Epworth Sleepiness Scale (ESS).
  Measurement will be taken prior to NIV initiation, 6 weeks post initiation and at follow up at 3 months.
Patients commencing on Non Invasive Ventilation (NIV); change in Exercise Capacity. | 3 months
  To demonstrate that the improvement in cardiac function and/or respiratory mechanics over time are associated with ongoing improvements in oxygenation by participants performing the Gate speed of 4 metres test prior to,during and after NIV initiation and at 6 weeks post initiation, and follow up at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Dr Steier, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Marino Dr Phil, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Foundation, London, United Kingdom

REFERENCES:
- See also: JTD publication — https://clinicaltrials.gov/ct2/show/NCT02699112?term=Steier&rank=3